CLINICAL TRIAL: NCT00387101
Title: Pivotal Study to Evaluate the Efficacy and Safety of Dermal-Living Skin Replacement (Dermal-LSR) in the Treatment of Chronic Diabetic Foot Ulcers
Brief Title: Efficacy and Safety Study in the Treatment of Chronic Diabetic Foot Ulcers
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low recruitment rate
Sponsor: ApoPharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RS03-2004
Record Dates: First submitted 2006-10-10; First posted 2006-10-12 (Estimated); Last update posted 2008-05-02 (Estimated); Status verified 2008-04

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetic Foot Ulcer; Diabetes Mellitus; Debridement; Dermal-LSR; Standard of Care
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus

INTERVENTIONS:
Device: Dermal - Living Skin Replacement (Dermal - LSR)

SUMMARY:
The purpose of this study is to determine the safety and efficacy of Dermal-LSR plus Standard of Care (SOC) for the treatment of diabetic foot ulcers (DFU)in comparison to the treatment to SOC alone.

DETAILED DESCRIPTION:
The study is a pivotal, prospective, randomized, controlled, open-label, multi-center study that will evaluate the effectiveness and safety of topically applied Dermal-LSR in chronic DFUs.

ELIGIBILITY:
Inclusion Criteria:

* Has signed a written informed consent prior to the first study intervention
* Is at least 18 and <85 years of age
* Has one or more diabetic foot ulcers on the target limb, with only one marked for the study (target ulcer). It must have the following characteristics:Plantar; Grade 2 per Curative Health Services Classification; Non-infected; Neuropathic; Non-malignant; At least 1.0-25cm^2 post-debridement; Present for at least 6 weeks
* Has Type I or II Diabetes Mellitus with an HBA1c between 6-10%
* Has a maximum fasting blood glucose level of 13.8 mmol/L
* An ankle-brachial systolic pressure index between 0.7 and 1.3
* If female and of childbearing potential has a negative serum pregnancy test and is neither breastfeeding or intending to become pregnant during the study
* Able and willing to attend the scheduled visits and comply with study procedures.

Exclusion Criteria:

* Known or suspected disease of the immune system
* Active or untreated malignancy or active, uncontrolled connective tissue disease
* Treatment with immunosuppressive or chemotherapeutic agents, radiotherapy or systemic corticosteroids less than 30 days before enrollment
* Presence of necrosis, purulence or sinus tracts that cannot be removed by debridement
* Has undergone revascularization procedure aimed at increasing blood flow in the treatment target limb < 4 weeks prior to enrollment
* Active febrile illness
* AST, ALT, ALP >3x the normal upper limit
* Serum Creatinine >2x the normal upper limit
* Osteomyelitis
* Active Charcot
* Use of any topical treatments other than SOC (standard of care)at the time of enrollment
* Enrollment in any investigational clinical trial within 30 days of the screening visit
* Known or suspected hypersensitivity to any study product components
* Recent or current history of alcohol or drug abuse
* Any condition, which in the opinion of the Investigator, would interfere with the evaluation of the study product or poses a health risk to the subject
* All site personnel directly affiliated with this study and their immediate families

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2006-02; Primary Completion 2007-09 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
To determine the efficacy and safety of Dermal-LSR plus Standard of Care (SOC) for the treatment of chronic diabetic foot ulcers in comparison to treatment with SOC alone.

CONTACTS AND LOCATIONS:
Overall Officials: Jason R Hanft, DPM, FAC FAS, Principal Investigator — Doctors Research Network, 7000 SW 62nd Avenue, Suite 310, South Miami, FL 33143; Hau Pham, DPM, Principal Investigator — Foot Care Vascular and Endovascular Specialists of Boston Medical Center, 732 Harrison Ave., 2nd Floor, Boston, MA 02118; Rodney Stuck, DPM, Principal Investigator — Hines VA Hospital, 5th and Roosevelt Rd., Building 200, 5th Floor, Room 501, Hines, IL 60141; Vickie Driver, DPM, Principal Investigator — National Center for Lower Limb Preservation, 8816 Dempster Street, Niles, Il 60714; Zevi Isseroff, DPM, Principal Investigator — North Shore Diabetic and Endocrine Associates, 3003 New Hyde Park Road Suite 201, New Hyde Park, NY, 11042; Lowell Weil, Jr., DPM, MBA, FAC FAS, Principal Investigator — Weil Foot and Ankle Institute, 1455 Golf Rd., Suite 110, Golf-River Professional Building, Des Plaines, IL 60016; Michal Drews, Principal Investigator — SPSK nr 2 im. H. Święcickiego AM Oddział Kliniczny Chirurgii Ogólnej Gastroenterologicznej i Endokrynologicznej ul. Przybyszewskiego 49; Henryk Komon, Principal Investigator — Centrum Medyczno-Diagnostyczne Sp. z o.o. ul. Piłsudskiego 49 08-110 Siedlce Poland; Krystyna Pilarska, Principal Investigator — SPWSZ w Szczecinie Klinika Endokrynologii, NadciśnieniaTętniczego i Chorób Przemiany Materii PAM ul. Arkońska 4 71-455 Szczecin; Malgorzata Wilczynska, Principal Investigator — NZOZ Centrum Opieki Diabetologiczno-Endokrynologicznej ul. Karola Miarki 6 50-306 Wrocław Poland; Joseph Cavorsi, M.D., Principal Investigator — Center for Advanced Wound Care 640 Walnut St., Suite 302 Reading, PA 19601; Roslyn R Isseroff, M.D., Principal Investigator — Veterans Affairs Northern Health Care System; Georgeanne Botek, DPM, Principal Investigator — The Learner Research Centre, Department of Orthopaedic Surgery. The Cleveland Clinic Foundation, 9500 Euclid Ave. A40, Cleveland, OH 44195,; Adam Landsman, DPM, PhD, Principal Investigator — Joslin-Beth Israel Deaconess Foot Center, Division of Podiatry, 185 Pilgrim Road, Boston, MA 02215; Jodi Walters, DPM, Principal Investigator — Southern Arizona Veterans Administration Health Care System, 3601 S. 6th Avenue (2-112), Tucson, AZ 85723; Martin Taubman, DPM, Principal Investigator — San Diego Research Center 4452 Park Boulevard Suite 210, San Diego, CA 92116
Locations (12):
- United States (12):
  - Southern Arizona Veterans Administration Health Care System, 3601 S. 6th Avenue (2-112), Tuscon, Arizona
  - Veterans Affairs Northern Health Care System, Sacramento VA Medical Center at Mather, Mather, California
  - San Diego Research Center 4452 Park Boulevard Suite 210, San Diego, San Diego, California
  - Doctors Research Network, South Miami, Florida
  - Weil Foot and Ankle Institute, Des Plaines, Illinois
  - Hines VA Hospital, Hines, Illinois
  - National Center for Lower Limb Preservation, Niles, Illinois
  - Foot Care Vascular and Endovascular Specialists of Boston Medical Center, Boston, Massachusetts
  - Joslin-Beth Israel Deaconess Foot Center, Division of Podiatry, 185 Pilgrim Road, Boston, Massachusetts
  - North Shore Diabetic and Endocrine Associates, New Hyde Park, New York
  - The Learner Research Centre, Department of Orthopaedic Surgery. The Cleveland Clinic Foundation, 9500 Euclid Ave. A40, Cleveland, Ohio
  - Center for Advanced Wound Care, Reading, Pennsylvania